CLINICAL TRIAL: NCT01768715
Title: Applicability of Liver Transplantation in Alcoholic Hepatitis
Brief Title: Liver Transplantation in Alcoholic Hepatitis
Acronym: SETH-HA
Status: Suspended | Type: Observational
Why Stopped: Low rate of recruitment (only one patient up to May 2014)
Sponsor: Sociedad Española de Trasplante Hepático (Network)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor
Other Study IDs: SETH-HA
Record Dates: First submitted 2012-12-29; First posted 2013-01-15 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic hepatitis; Liver transplantation; Survival; Alcoholism
MeSH Terms: conditions — Hepatitis, Alcoholic; Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Good response: Patients with severe alcoholic hepatitis and good response to therapy.
- Non transplant candidates: Patients with severe alcoholic hepatitis and poor response to therapy, that are not candidates to transplantation, according to the specified criteria.
- Transplant candidates: Patients with severe alcoholic hepatitis and poor response to therapy, that are candidates to transplantation, according to the specified criteria.

SUMMARY:
Patients with alcoholic hepatitis non-responsive to steroids have a poor prognosis. Recently a French-Belgian prospective study has obtained good results (acceptable survival with a low rate of alcohol recidivism).

The hypothesis of the present study is that carefully selected Spanish patients with alcoholic hepatitis that do not respond to steroid therapy may have a good survival if they receive a liver transplant. The expected rate of alcohol recidivism in such a selected population will be low.

DETAILED DESCRIPTION:
This is a open prospective multicenter study. Nineteen liver transplant units in Spain will take part in it.

Inclusion criteria for patients:

1. Diagnosis of alcoholic hepatitis (liver biopsy will be advisable).
2. First episode of clinical decompensation of alcoholic liver disease (defined as jaundice, variceal bleeding, ascites or portal-systemic encephalopathy).
3. Absence of a high risk of alcoholic recidivism (according to De Gottardi, et al).
4. Severe alcoholic hepatitis (ABIC score > 6.71)
5. Informed consent

Exclusion criteria :

1. Age over 65 years.
2. Hepatitis B or C or HIV infections.
3. Uncontrolled bacterial infection
4. Other liver diseases, such as alpha-1-antitrypsin deficiency, primary biliary cirrhosis, ...
5. Morbid obesity (BMI > 35 kg/m2)
6. Major uncontrolled psychiatric disease
7. Drug addiction (excluding tobacco) in the last two years.
8. Absence of informed consent.
9. Acute-on-chronic liver disease.
10. Paracetamol consumption over 10 grams in the last week.

Criteria for liver transplantation.

1. Absence of response to steroid therapy (Lille score ≥ 0.45 7 days after initiation of steroid therapy).
2. Adequate social and familiar environment.
3. Complete agreement in the medical staff about the candidate to transplantation.
4. Absence of bacterial or fungal infection.

Three groups of patients will be formed:

Group 1. Patients with severe alcoholic hepatitis and good response to therapy. Group 2. Patients with severe alcoholic hepatitis and poor response to therapy, that are not candidates to transplantation.

Group 3. Patients with severe alcoholic hepatitis and poor response to therapy, that are candidates to transplantation.

A complete follow-up of the patients would be extended to five years. The survival of these three groups will be compared. Survival of liver transplant recipients should also be compared with survival of other liver transplant recipients.

Alcohol recidivism should also be studied in all the patients of the study. Sample size estimation: According to the data published by Mathurin et al, 28 patients treated with liver transplantation and 28 non-transplanted patients with severe alcoholic hepatitis should be necessary.

Interim analysis after every 10 transplanted patients should be performed. The study will be interrupted if the differences in the survivals between groups 2 and 3 reaches a significance of 0.01. In case this significance is not reached the inclusion of patients should end when 40 patients are transplanted. This sample size is estimated to be reached in 18-24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of alcoholic hepatitis (liver biopsy will be advisable).
2. First episode of clinical decompensation of alcoholic liver disease (defined as jaundice, variceal bleeding, ascites or portal-systemic encephalopathy).
3. Absence of a high risk of alcoholic recidivism (according to De Gottardi, et al).
4. Severe alcoholic hepatitis (ABIC score > 6.71)
5. Informed consent

Exclusion Criteria:

1. Age over 65 years.
2. Hepatitis B or C or HIV infections.
3. Uncontrolled bacterial infection
4. Other liver diseases, such as alpha-1-antitrypsin deficiency, primary biliary cirrhosis, ...
5. Morbid obesity (BMI > 35 kg/m2)
6. Major uncontrolled psychiatric disease
7. Drug addiction (excluding tobacco) in the last two years.
8. Absence of informed consent.
9. Acute-on-chronic liver disease.
10. Paracetamol consumption over 10 grams in the last week.

Criteria for liver transplantation.

1. Absence of response to steroid therapy (Lille score ≥ 0.45 7 days after initiation of steroid therapy).
2. Adequate social and familiar environment.
3. Complete agreement in the medical staff about the candidate to transplantation.
4. Absence of bacterial or fungal infection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with alcoholic hepatitis participating in this trial are going to be selected from patients admitted to the hospital (from the emergency department or referred from other hospital)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate survival of patients with severe alcoholic hepatitis non responsive to therapy after liver transplantation | 1 year after the diagnosis of alcoholic hepatitis
  The survival of patients transplanted with alcoholic hepatitis is going to be compared with the survival of patients with alcoholic hepatitis that are not considered adequate for liver transplantation

SECONDARY OUTCOMES:
Evaluate the applicability of liver transplantation in patients with alcoholic hepatitis non responsive to steroid therapy | 1 year
  The applicability of liver transplantation is defined as the ratio between the number of patients transplanted for alcoholic hepatitis and the number of patients with severe alcoholic hepatitis that do not respond to steroid therapy.
Evaluate the mortality in waiting list for transplantation of patients with alcoholic hepatitis unresponsive to steroid therapy | 1 year
  Proportion of patients who are accepted as candidates for liver transplantation who die before transplantation.
Evaluate the rate of alcohol recidivism after liver transplantation for alcoholic hepatitis | 1, 2, 3, 4 and 5 years
  Proportion of patients transplanted for alcoholic hepatitis that have a recurrence in alcohol consumption
Evaluate survival of patients with alcoholic hepatitis after liver transplantation. | 2, 3, 4 and 5 years after the diagnosis of alcoholic hepatitis
  The survival of patients transplanted with alcoholic hepatitis is going to be compared with the survival of patients with alcoholic hepatitis that are not considered adequate for liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Herrero, MD, Study Chair — Clinica Universidad de Navarra; Santiago Tome, MD, Study Chair — Complejo Hospitalario Universitario de Santiago; Ignacio Gonzalez-Pinto, MD, Study Chair — Hospital Central de Asturias
Locations (17):
- Spain (17):
  - Hospital Vall d'Hebrón, Barcelona, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Virgen de la Nieves, Granada, Granada
  - Complejo Hospitalario Universitario de la Coruña, A Coruña, La Coruña
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Carlos Haya, Málaga, Málaga
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Virgen del Rocío, Seville, Sevilla
  - Hospital La Fe, Valencia, Valencia
  - Hospital Río Hortega, Valladolid, Valladolid
  - Hospital Lozano Blesa, Zaragoza, Zaragoza

REFERENCES:
- [Background] Dominguez M, Rincon D, Abraldes JG, Miquel R, Colmenero J, Bellot P, Garcia-Pagan JC, Fernandez R, Moreno M, Banares R, Arroyo V, Caballeria J, Gines P, Bataller R. A new scoring system for prognostic stratification of patients with alcoholic hepatitis. Am J Gastroenterol. 2008 Nov;103(11):2747-56. doi: 10.1111/j.1572-0241.2008.02104.x. Epub 2008 Aug 21. PMID 18721242
- [Background] Tome S, Martinez-Rey C, Gonzalez-Quintela A, Gude F, Brage A, Otero E, Abdulkader I, Forteza J, Bustamante M, Varo E. Influence of superimposed alcoholic hepatitis on the outcome of liver transplantation for end-stage alcoholic liver disease. J Hepatol. 2002 Jun;36(6):793-8. doi: 10.1016/s0168-8278(02)00047-8. PMID 12044530
- [Background] Wells JT, Said A, Agni R, Tome S, Hughes S, Dureja P, Lucey MR. The impact of acute alcoholic hepatitis in the explanted recipient liver on outcome after liver transplantation. Liver Transpl. 2007 Dec;13(12):1728-35. doi: 10.1002/lt.21298. PMID 18044757
- [Background] Mathurin P, Moreno C, Samuel D, Dumortier J, Salleron J, Durand F, Castel H, Duhamel A, Pageaux GP, Leroy V, Dharancy S, Louvet A, Boleslawski E, Lucidi V, Gustot T, Francoz C, Letoublon C, Castaing D, Belghiti J, Donckier V, Pruvot FR, Duclos-Vallee JC. Early liver transplantation for severe alcoholic hepatitis. N Engl J Med. 2011 Nov 10;365(19):1790-800. doi: 10.1056/NEJMoa1105703. PMID 22070476